CLINICAL TRIAL: NCT02361658
Title: Ultrasonographic Assessment of the Optic Nerve Sheath Diameter During Variations in PetCO2 and Controlled Internal Jugular Venous Occlusion: A Volunteer Study
Brief Title: Optic Nerve Sheath Diameter (ONSD) With the Raised PCO2 and Internal Jugular Venous Occlusion
Status: Completed | Type: Observational
Sponsor: Lashmi Venkatraghavan (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor-Investigator, Lashmi Venkatraghavan, Assistant Professor, Department of Anesthesia, Toronto Western Hospital, Toronto, Canada, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Other Study IDs: UHN REB # 14-8014
Record Dates: First submitted 2015-02-03; First posted 2015-02-12 (Estimated); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Elevated Intracranial Pressure (ICP)
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasonographic of the optic nerve sheath diameter — On both eyes of all subjects in supine position by two investigators.
Other: RespirAct™ — Carbon dioxide Manipulation by RespirAct™ sequential gas delivery breathing circuit at each CO2 levels (normocapnia, Hypercapnia I and II and hypocapnia).
Other: Neck collar — Internal jugular compression using a Neck collar will be applied at each CO2 levels (normocapnia, Hypercapnia I and II and hypocapnia) and ONSD measurements will be done before and after the collar.

SUMMARY:
Monitoring the ICP is the most important aspect of the management of these patients. Recently, transorbital ultrasonography has gained popularity as a noninvasive bedside exam that has been shown to be useful in the diagnosis of raised ICP by evaluating the change in the optic nerve sheath diameter (ONSD). Transorbital ultrasonographic measurement of ONSD appears to be a noninvasive, relatively inexpensive bedside examination for the diagnosis of raised ICP. The investigators aimed to determine the changes in ONSD with acute controlled changes in ICP in healthy volunteers. The controlled changes in ICP will be produced by manipulating the PCO2 with the use of Respiract and jugular venous compression with the use of custom made neck collar.

DETAILED DESCRIPTION:
Elevated intracranial pressure (ICP) is a common and potentially life threatening condition arising from a variety of pathological conditions including traumatic brain injury (TBI), intracranial hemorrhage, subarachnoid hemorrhage and brain tumors. Monitoring the ICP is the most important aspect of the management of these patients. Recently, transorbital ultrasonography has gained popularity as a noninvasive bedside exam that has been shown to be useful in the diagnosis of raised ICP by evaluating the change in the optic nerve sheath diameter (ONSD). Transorbital ultrasonographic measurement of ONSD appears to be a noninvasive, relatively inexpensive bedside examination for the diagnosis of raised ICP. The investigators aimed to determine the changes in ONSD with acute controlled changes in ICP in healthy volunteers. The controlled changes in ICP will be produced by manipulating the PCO2 with the use of Respiract and jugular venous compression with the use of custom made neck collar.

ELIGIBILITY:
Inclusion Criteria:

Adult healthy volunteers who are above the age of 18 ASA 1 Body mass index (BMI) less than and equal to 35 Neurologically normal subjects with no symptoms other than occasional non-severe headache

Exclusion Criteria:

BMI above 35 Lack of informed consent Language barrier Medical students and/or anesthesia residents going through the department as part of their rotation Pregnancy Frequent migraine headache

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lashmi Venkatraghavan, MD, Principal Investigator — Assistant Professor, Toronto Western Hospital, University Health Network
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult healthy volunteers who are above the age of 18 ASA 1 Body mass index (BMI) less than and equal to 35 Neurologically normal subjects with no symptoms other than occasional non-severe headache
Groups:
- Ultrasonographic of the Optic Nerve Sheath Diameter: Use transorbital ultrasound to evaluate ONSD changes in patients with intracranial pathology and to compare the changes in the ONSD before and after surgical intervention as well as between patients with and without clinical or radiological signs of increased ICP
Period: Overall Study
Arm/Group | Ultrasonographic of the Optic Nerve Sheath Diameter
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ultrasonographic of the Optic Nerve Sheath Diameter
Number analyzed (Participants) | 100
Age, Customized [Count of Participants; unit: Participants]
  Participants | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 100
Intracranial pathology scheduled for elective or emergency surgery [Count of Participants; unit: Participants] | 100

OUTCOME MEASURES:

1. Primary Outcome: Changes in ONSD in mm With Changes in ICP in Healthy Volunteers.
Description: Transorbital ultrasound will be used for measuring the changes in ONSD. The controlled changes in ICP will be produced by manipulating the PCO2 with the use of Respiract and jugular venous compression with the use of custom made neck collar.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Ultrasonographic of the Optic Nerve Sheath Diameter: Transorbital ultrasound will be used for measuring the changes in ONSD. The controlled changes in ICP will be produced by manipulating the PCO2 with the use of Respiract and jugular venous compression with the use of custom made neck collar.
Arm/Group | Ultrasonographic of the Optic Nerve Sheath Diameter
Number analyzed (Participants) | 100
mm | 4.2 (0.7)

ADVERSE EVENTS:
Time Frame: one day to 8 weeks
Description: Ultrasound Gel can be cold on contact with skin.
Arm/Group | Ultrasonographic of the Optic Nerve Sheath Diameter
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT02361658/Prot_SAP_000.pdf